CLINICAL TRIAL: NCT04225585
Title: Improving Well-Being for Individuals With Persistent Pain After Surgery for Breast Cancer, Lobular Carcinoma in Situ, or Ductal Carcinoma in Situ: A Randomized Clinical Trial That Compares Three Behavioral Intervention Strategies and Examines Psychological Factors as Drivers of the Continuing Burden of Persistent Pain
Brief Title: Well-Being After Breast Cancer Surgery
Acronym: WB ABCs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00104214
Record Dates: First submitted 2020-01-03; First posted 2020-01-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Coping Skills Training for Persistent Post-Surgical Pain; General Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study staff conducting assessments will be blind to group assignment. To maintain blinding, we will use the following approaches: 1) all study staff will be trained on the importance of blinding and study procedures to maintain blinding; 2) participants will be provided with the rationale and instructions not to disclose their group assignment; 3) the study staff who conduct post-intervention assessments will not be given information about group assignment prior to the assessment; and 4) if a breach occurs, it will be documented and the participant will complete their assessment with a new assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coping Skills Training for Persistent Post-Surgical Pain (Experimental): novel pain coping skills training intervention designed specifically for people with persistent pain (PP) following breast cancer surgery
  Interventions: Behavioral: CST-PSP
- General health education with a coach (Active Comparator): general health education intervention
  Interventions: Behavioral: General health education
- Self-guided health education (Active Comparator): general health education intervention
  Interventions: Behavioral: General health education

INTERVENTIONS:
Behavioral: CST-PSP — skills training and experiential learning exercises
  Other Names: Coping Skills Training for Persistent Post-Surgical Pain
  Arms: Coping Skills Training for Persistent Post-Surgical Pain
Behavioral: General health education — general health education intervention that focuses on improving overall health
  Arms: General health education with a coach; Self-guided health education

SUMMARY:
The purpose of this study is to compare the benefits of skills training and health education interventions designed specifically to increase the well-being of people with persistent pain after breast surgery for lobular carcinoma in situ (LCIS), ductal carcinoma in situ (DCIS), or invasive breast cancer, and to examine the roles of psychological and physiological variables as modifiable contributors to the continuing burden of persistent pain.

DETAILED DESCRIPTION:
Persistent pain following breast surgery for lobular carcinoma in situ (LCIS), ductal carcinoma in situ (DCIS), or invasive breast cancer is increasingly recognized as an important clinical and public health issue due to the large number of women affected, the powerful negative impact that persistent pain has on emotional and physical functioning and its financial costs. Most of the more than a quarter of a million women newly diagnosed with breast cancer in the U.S. this year will undergo surgery as a part of curative treatment. The prevalence of persistent pain following surgical removal of the affected breast (mastectomy) or more limited surgeries (lumpectomy) is high, ranging from 25-60% across studies. Unlike acute post-operative pain, which is a normal response to surgical trauma, persistent pain at or near the surgical site has an uncertain multifaceted etiology, and no satisfactory pharmacological treatment. A critical question is whether key pain-related psychosocial factors are drivers of the continuing burden of persistent pain, and whether they could be ameliorated by non-pharmacological intervention. The research planned under this award will provide a first critical test of the hypothesized driving role of pain catastrophizing in persistent pain after breast surgery. It also will explore the role of two other key psychosocial variables that may contribute to the burden associated with persistent pain after breast cancer surgery: self-efficacy for engaging in valued activities and psychological inflexibility. We have developed, manualized, and pilot tested a pain coping skills training intervention that specifically targets the needs of women with persistent pain following breast cancer surgery (CST-PSP) and aims to reduce pain catastrophizing, increase self-efficacy for engaging in valued activities, and increase psychological flexibility. We propose a multiple-site, randomized clinical trial to evaluate the efficacy of the CST-PSP intervention, as well as a health education intervention. The study will be conducted in diverse oncology clinics affiliated with Duke University/Duke Cancer Network and the University of Pittsburgh/UPMC Hillman Cancer Center. Participants (N=316) will be randomized to either receive: 1) CST-PSP, 2) health education with an interventionist, or 3) self-guided health education . Participants will complete assessments pre-intervention and at 3 months (post-intervention), 6 months follow-up, and 12 months follow-up. Study aims are: Aim 1: Examine the impact of intervention programs on persistent post-surgical pain severity and interference (i.e., PEG score), emotional distress (anxiety and depression), and cancer-specific distress. Aim 2: Investigate the impact of intervention programs on pain catastrophizing, pain self-efficacy, and psychological inflexibility, and evaluate these variables as possible mediators of the intervention benefits. Aim 3: Evaluate the impact of intervention programs on pain sensitivity and central sensitization, and explore whether changes in these variables mediate group differences in pain severity and interference.

ELIGIBILITY:
Inclusion Criteria:

* prior diagnosis of Stage 0 to III breast cancer, DCIS or LCiS
* received first breast cancer surgery (total or partial mastectomy, lumpectomy) at least 3 months ago
* reports score of ≥3 in the past month on the 0 to 10 breast pain severity and/or interference scale
* able to speak and read English
* able to provide meaningful consent

Exclusion Criteria:

* <18 years of age
* hearing impairment that limits use of videoconferencing for intervention sessions
* cognitive impairment that is documented in the medical record or results in being unable to provide meaningful consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in PEG Pain Severity and Interference | Baseline, 3 months, 6 months, 12 months
  Persistent post-surgical pain burden 3-item measure: average pain intensity (P); interference with enjoyment in life (E); interference with general activity (G)

SECONDARY OUTCOMES:
Change in emotional distress: Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Baseline, 3 months, 6 months, 12 months
  Composite score of 8-item assessment of depressive symptoms over the past two weeks and 7-item assessment of symptoms of anxiety over the past two weeks
Change in pain catastrophizing: Pain Catastrophizing Scale (PCS) | Baseline, 3 months, 6 months, 12 months
  13-item assessment of the degree to which participants experience catastrophic thinking during painful experiences
Change in Central sensitization: Central Sensitization Inventory (CSI) | Baseline, 3 months, 6 months, 12 months
  25-item questionnaire designed to measure hypersensitivity to senses and signs of central sensitization
Change in Central sensitization: Temporal summation | Baseline, 6 months, 12 months
  Designed to measure central pain mediation using weighted pinprick probes

OTHER OUTCOMES:
Change in cancer-specific distress: Impact of Event Scale (IES) | Baseline, 3 months, 6 months, 12 months
  15-item measure of intrusive and avoidant cognition regarding breast cancer during the past week
Change in psychological inflexibility: Acceptance and Action Questionnaire (AAQ-II) | Baseline, 3 months, 6 months, 12 months
  7-item questionnaire designed to measure psychological inflexibility
Change in self-efficacy: Chronic Pain Self-Efficacy Scale: Function Self-Efficacy Subscale (FSE) | Baseline, 3 months, 6 months, 12 months
  9-item questionnaire designed to measure chronic pain patients' perceived self-efficacy for engaging in activities
Change in Pain sensitivity: Pressure pain thresholds | Baseline, 6 months, 12 months
  Designed to measure central hyperexcitability using a digital pressure algometer measured pressure that is first perceived as painful and recorded in kg
Change in Pain sensitivity: Mechanical cutaneous pain thresholds | Baseline, 6 months, 12 months
  Assessed using weighted pinprick probes with standard stimulus intensities (8, 16, 32, 64, 128, 256, and 512 mN) and contact areas (tip diameter 0.20 mm). Stimuli are applied to the middle phalanx of digit 3, beginning with the lowest-force stimulator until the suprathreshold value is reached. The direction of the testing is then changed toward lower stimulus intensities until the probe stimulation is perceived as 'touch' only (sub-threshold value). Testing then directs again toward higher intensities, until 5 suprathreshold and 5 subthreshold values have been recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Shelby, PhD, Principal Investigator — Duke University; Dana Bovbjerg, PhD, Principal Investigator — University of Pittsburgh Medical Center
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stalls JM, Bovbjerg DH, Somers TJ, Plumb Vilardaga JC, Kimmick GG, McAuliffe PF, Keefe FJ, Posluszny DM, Sullivan MJL, Erkanli A, Reed SD, Sutton L, Owen L, Massa L, Shelby RA. Improving well-being for individuals with persistent pain after surgery for breast cancer, lobular carcinoma in situ, or ductal carcinoma in situ: A randomized clinical trial. Contemp Clin Trials. 2022 Nov;122:106934. doi: 10.1016/j.cct.2022.106934. Epub 2022 Sep 21. PMID 36152791

DOCUMENTS (1):
  • Informed Consent Form (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT04225585/ICF_000.pdf